CLINICAL TRIAL: NCT04661319
Title: Impact of Video Editing Training for Novice Trainees in Laparoscopic Cholecystectomy; a Multicenter, Randomized, Controlled Trial
Brief Title: Impact of Video Editing Training for Novice Trainees in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Seoul-10
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Gallstone; Colic
Keywords: video editing training; laparoscopic cholecystectomy; novice trainees
MeSH Terms: conditions — Gallstones; Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video editing training group (Experimental): - inclusion criteria
  1. trainees in general surgery
  2. No experience of laparoscopic cholecystectomy
  3. Less than 5 experiences of laparoscopic surgery
  4. Uncomplicated symptomatic gallstone disease
  The experimental group received video editing training
  Interventions: Procedure: video editing training
- traditional training group (Experimental): - inclusion criteria
  1. trainees in general surgery
  2. No experience of laparoscopic cholecystectomy
  3. Less than 5 experiences of laparoscopic surgery
  4. Uncomplicated symptomatic gallstone disease
  The control group received tradtional training
  Interventions: Procedure: video editing training

INTERVENTIONS:
Procedure: video editing training — 1. The subject's preoperative residency year, instrument experience, open surgery experience, laparoscopic surgery experience, and preoperative instrument proficiency are evaluated.
  2. Basic anatomical and scientific education for laparoscopic cholecystectomy, practice laparoscopic instruments for at least 30 minutes every other week, and observe 3 cases of laparoscopic cholecystectomy.
  3. Select a random experimental group.
  4. For each selected group, 3 cases of surgical observation or 3 cases of video editing are performed.
  5. Both groups operated on 10 cases, and both groups were discharged from the hospital after undergoing the same recovery procedure after the same operation.

SUMMARY:
Surgical practice training often suffers from poor educational efficiency due to the technical difficulties of the cases, the lack of resources and the cases in the operating room. The video editing training method is not included in the standard surgical training, but it has the advantage of reducing trial and error and errors during surgery, simplifying training time, and cost-effective. Investigators analyzed whether the video editing teaching method has effective value for trainees compared to the traditional teaching method.

The primary purpose of the study is the trainee's learning achievement in terms of surgical skills. Learning achievement is measured as the difference in pre- and post-educational test scores (The Global Operative Assessment of Laparoscopic Skills (GOALS)) to compare the difference in achievement.

The secondary objective of the study was to evaluate the satisfaction with the video editing method as an educational method by conducting a questionnaire survey to all the trainees participating in the study. In addition, the degree of postoperative pain, postoperative hospitalization period, postoperative readmission and the need for additional procedures were compared and analyzed.

DETAILED DESCRIPTION:
1. background Traditional education teaches surgery in a one-on-one apprenticeship of surgeons and practitioners, in which the surgeon learns to perform surgical operations under the supervision of a qualified surgeon. The supervisor surgeon instructs the trainee and, if necessary, temporarily takes over the procedure to show the difficult steps. Today, a proven educational platform has been established to prevent the risk of patients being exposed to the early learning curve, allowing trainees to sufficiently hone their basic skills in open and laparoscopic surgery.

   Laparoscopic surgery requires complex techniques and techniques that are not used in open surgery. Laparoscopic instruments provide limited haptic feedback, lack of freedom, and video monitors that provide a two-dimensional projection of the operating room impair depth perception, making surgery more difficult. Therefore, surgeons must master these technical challenges before performing laparoscopic procedures properly and safely.

   Animal model training and cadaver training are very useful, but have the disadvantages of being small in number and expensive to use. On the other hand, books, the Internet, and educational videos have the advantage of being able to provide important basic knowledge about disease and surgical treatment, but the most important factor in training specific surgical procedures is from the trainee side to the real patient together with an experienced surgeon Since it is a practical training for Korea, the teaching method still used is the apprenticeship method. The main drawback of this traditional approach is that the trainee or supervising surgeon can only perform the step once per operation. When the supervisor takes over, the memories of training with the trainee who have to wait for the next task to be performed are lost.

   Therefore, investigators devised a new training method called surgical video editing in order to minimize the frequency of supervisor intervention and maximize the actual surgical practice time of the trainee. This method is used by the trainee himself to review the surgical process, Since the essential skills can be recalled and learned, it can have the effect that the trainee can easily learn the surgery during the actual surgery.
2. Target disease : Patients with uncomplicated symptomatic gallstone disease who are scheduled operation
3. Selection criteria, exclusion criteria, target number of subjects

   1. inclusion criteria

      1. trainees in general surgery
      2. No experience of laparoscopic cholecystectomy
      3. Less than 5 experiences of laparoscopic surgery
      4. Uncomplicated symptomatic gallstone disease
   2. Exclusion Criteria

      1. Experience with laparoscopic cholecystectomy.
      2. More than 5 experiences of laparoscopic surgery
   3. Target number and evidence In the existing literature, it was assumed that the difference between the video editing group and the control group in the primary result was 20% or more. This difference was assumed to be a 2-sided confidence level of 95% with a power of two-sided significance level α = 0.2 and power 80%, and 45 subjects were assigned to each group considering the dropout rate of 10%.
   4. Random allocation schedule and operation Randomization was assigned using block randomization without stratification, and in order to maintain unpredictability, which is the basic principle of randomization, the randomization table will be completed by applying a block size of 2 or 4 or 6. .

   The allocation envelope in which the randomization number and allocation group are recorded is made of opaque material so that it can be blinded, and it is kept sealed until randomization is performed for each subject.

   The person in charge of the clinical trial or the person in charge of the clinical trial finally confirms the criteria for exclusion, and if the subject is suitable, assigns a random assignment number and keeps it in the assignment bag. Afterwards, the study nurse unseals the assignment bag with the assignment number and conducts D education in the administration group assigned to the subject according to each random assignment number. The research nurse must record the release information (release date and release person) immediately upon release of the sealing of the assignment envelope, and the random assignment envelope that has already been released can be re-assigned to another subject even if the subject has withdrawn consent will not be.
4. Clinical test method (administration/dosage, administration/use method, administration/use period, combination therapy, etc.) A. study design : Prospective multicenter randomized controlled trial B. Describe the treatment for the experimental group / control group

   1. Clinical trial flow

      1. The subject's preoperative residency year, instrument experience, open surgery experience, laparoscopic surgery experience, and preoperative instrument proficiency are evaluated.
      2. Basic anatomical and scientific education for laparoscopic cholecystectomy, practice laparoscopic instruments for at least 30 minutes every other week, and observe 3 cases of laparoscopic cholecystectomy.
      3. Select a random experimental group.
      4. For each selected group, 3 cases of surgical observation or 3 cases of video editing are performed.

         * The person in charge of the clinical trial or the person in charge of the clinical trial finally confirms the criteria for exclusion from selection, and if the subject is suitable, assigns a random assignment number and keeps it in the assignment bag. After that, the research nurse receives the assignment bag with the assignment number and unseals the assignment bag to proceed with the training method according to the assigned group assigned to the subject according to each random assignment number.
      5. Both groups operated on 10 cases, and both groups were discharged from the hospital after undergoing the same recovery procedure after the same operation.
      6. Patients undergo a hematological test, blood chemistry test, urine test, coagulation test, and chest x-ray on the first day after surgery. (Examination and treatment are performed according to the Clinical Pathway of the current gallbladder surgery-clinical practice guidelines-)
      7. If there are no specifics, patients should start with a liquid meal in the morning of the first day after surgery.
      8. Patients are discharged from the hospital on the 2nd day after surgery if there are no specifics.
      9. Follow-up of complications during hospitalization and after discharge of patients.
   2. Surgery method

      1. Start the operation under general anesthesia.
      2. Install a trocar of 10mm on the navel, 5mm below the knuckle, and 5mm on the right upper abdomen.
      3. Relief surgery is performed using CO2 gas in the abdominal cavity. -The back pressure through CO2 gas is maintained at 12mmHg/and 2L/min.
      4. Start dissection from Calot's triangle and proceed with the surgery using the retrograde cholecystectomy method. -The gallbladder duct is ligated with a 10mm clip and the gallbladder artery is also ligated with a 10mm clip. -If the gallbladder duct is ligated unstable, perform ligation through an endoloop. -After ligation, the gallbladder is detached from the liver.
      5. Wash the surgical site.
      6. Put the exfoliated gallbladder in a laparoscopic pocket and discharge it through the navel.
      7. Remove the trocar, suture the skin, and finish the operation.
   3. Discharge principle

      1. When hematologically stable and vital signs are stable
      2. When the patient's condition is stable by proceeding to a normal liquid diet
5. Observation variables/clinical test item and observation test method A. Observation item

   1. Pre-test investigation Before entering the clinical trial, the following matters are checked through interviews, chart checks, and questions about the subject's background (demographic information), and recorded in the case record.

      1. Background check: Subject's initials, date of birth, gender, residency year, instrument experience, open surgery experience, laparoscopic surgery experience, preoperative instrument skill evaluation
      2. Patients undergoing surgery: history, sex, age, diagnosis,
   2. Examination of surgical technique before operation

      ① Laparoscopic cholecystectomy The surgical image is viewed, and the anatomical structure and surgical process in the image, and the necessary technical areas (correct placement of trocar, carrot triangle structure, related anatomy, clip placement and resection structure) are evaluated and scored.
      * Basic Laparoscopic Skills Assessment: The Global Operative Assessment of Laparoscopic Skills (GOALS)
   3. Examination of surgical technique

      * The Global Operative Assessment of Laparoscopic Skills (GOALS) and technical rating scale (TRS) by viewing images of two groups of laparoscopic cholecystectomy

        * In case of intervention of supervisor during surgery: 0.5 point deduction for verbal intervention and 1 point deduction for behavioral intervention.
   4. Subject evaluation

      * Evaluating the anatomical structure during surgery and how difficult the surgical procedure was: a score of 10

        * Confidence in overall operation progress: evaluated with a score of 10 ③ Value of surgical observation and video editing on the progress of the surgery: evaluated as a score of 10
   5. Patients who underwent surgery

      * Hospital stay period after surgery, hematological test the day after surgery, blood chemistry test, urine test, blood coagulation test

        * Surgical site infection

          - Check at each patient visit. If there is redness, hot sensation, or abscess at the site of trocar insertion, it is defined as a superficial surgical site infection.

          - If there is fluid retention and abscess around the surgical site in the abdominal cavity, it is defined as a deep surgical site infection.
          * Distant infection : : Respiratory and urinary system infections and bacteremia or lymphatic inflammation ③ Check for bile leakage.
          * Groups with drainage pipes are identified through the drainage pattern. In the group without drainage tube, selective radiological follow-up (CT, sonogram, MRCP) was performed in cases of epigastric pain, indigestion, fever, and jaundice after surgery.
   6. Surgery time, blood loss description.
   7. Describe post-operative complications (other than those described above).
6. Predicted side effects and precautions for use : none
7. Criteria for stopping/dropping of the study When the following occurs, the test should be stopped, and the reason and findings of the interruption should be recorded in the case record.

<!-- -->

1. In the case that a patient's life-threatening side effect is expressed after surgery, and the investigator determines that it is necessary to stop
2. In case the subject refuses or withdraws consent after the start of the test
3. If it is determined that it is inappropriate as a target patient after starting the test
4. In the case of receiving training that can affect the improvement of surgical skills, such as other cadeveric practice, without the permission of the test manager after the start of the test
5. When it is judged that it is impossible to conduct an inspection or investigation after the start of the test due to the circumstances of the subject
6. In case the test manager determines that it is necessary to stop the test after the initiation of the test because it is life-threatening or the effect is manifested during surgery.

8. Effect evaluation criteria, evaluation method and interpretation method (statistical analysis method)

1. Analysis of efficacy variables

   - Analysis of primary efficacy variables.

   : Measured by the difference between the trainee's pre- and post-educational test scores (The Global Operative Assessment of Laparoscopic Skills, GOALS), and tested using the student's t-test or wilcoxn's rank sum test according to the satisfaction of the normal distribution assumption, Descriptive statistics (mean, standard deviation, median, minimum, maximum) are presented. In addition, the difference between the two groups' test scores (test group-control group) is presented as the mean and 95% confidence interval, and it can be confirmed that there was a learning effect when the difference in test score improvement between the two groups was 20% or more.
2. Analysis of secondary efficacy variables For categorical variables for hospital stay, operation time, and complication data obtained as secondary endpoints, n (%) is presented, and the difference in ratio between the two groups is tested using Chi-square or Fisher's exact test. In the case of continuous variables, the mean, standard deviation, median, minimum, and maximum values are presented, and normality tests are performed to test with Student's t-test for normal distribution, and Wilcoxon rank-sum test for nonnormal distribution. The investigators will test the difference between the two groups. For all statistical analysis, SPSS version 21.0 will be used, and those below the significance level of 0.05 will be judged as statistically significant.
3. Analysis target group

   1. intention to treat analysis group Randomization is performed only when the selection criteria described above are met, and all randomized subjects are to be included in the statistical analysis.
   2. per protocol analysis group The per protocol analysis group is defined as a trainee whose training has ended after receiving random assignments and assessed test scores.
4. How to deal with missing values This study is a prospective study, and it is expected that there will be no missing values of the primary or secondary endpoints during the experiment period. However, if missing values occur, the missing values should be substituted with the average value.
5. How to handle compliance Since the intervention applied in this study is an intervention performed during surgery while the patient is under general anesthesia, there will be no difference in treatment compliance. In addition, postoperative chest radiography and pain assessment have been previously included in the clinical pathway of laparoscopic cholecystectomy, so there is no difference in treatment compliance.

   9. Safety evaluation criteria including side effects, evaluation methods and reporting methods In the event of adverse reactions and side effects after surgery, subjects are educated to report to the researcher, and the occurrence of adverse reactions is checked and recorded at each visit, and symptoms, time of appearance, duration, degree of adverse reactions, and causal relationship with test drugs Are recorded in the case record. In the event of serious adverse reactions or unexpected problems, the lead researcher should report to the IRB.

   10. Rules for compensation for victims Laparoscopic cholecystectomy is a safe operation with extremely low risk of surgery. Also, there are basically no additional risks that accompany the study. Since antibiotics are drugs that have been used previously, there is no additional occurrence other than known complications. If participants get an injury or illness by participating in this study, medical treatment will be provided. The investigators will provide participants with a quick diagnosis and treatment if necessary through a referral for consultation with a medical professional related to the relevant clinical symptoms or signs.

   11. preparation for the safety protection of subjects 19.1 Clinical trial agency The head of the conducting institution shall make every effort to protect the safety of the subjects by equipping them with the necessary facilities and specialized personnel for conducting the relevant clinical trial step by step so that the clinical trial can proceed properly as specified in this study protocol. The person in charge of the clinical trial must fully understand the side effects and cautions specified in this plan in advance, and if any serious side effects occur during the study, immediately stop the clinical trial of the patient, take appropriate measures, and notify the relevant review committee.

19.2 Approval and revision of clinical trial protocol In the case of obtaining approval of a clinical trial or intending to perform a modified clinical trial, approval is obtained from the Institutional Review Board.

19.3 Familiarity with the research plan The study manager and the person in charge accurately analyze and understand the research plan, and actively respond to the subject's problems.

19.4 Clinical Trial Consent Before entering the clinical study, after explaining all the contents and safety of the test to the subject, the subject himself/herself voluntarily obtains consent to participate in this study and enters the study.

19.5 Selecting the correct subject Prior to this study, the suitability of the subject is thoroughly evaluated. 19.6 Subject's Confidentiality Records that can identify the subject will be kept confidential, and even if the results of the clinical trial are published, the subject's identity will be kept confidential.

All documents related to clinical trials, such as case records, should be recorded and classified with the subject identification code (usually the patient's initial), not the patient name.

19.7 Clinical trial drug management : None. 19.8 Action in case of adverse reaction In the event of an adverse reaction, it is managed to receive the necessary examination and treatment from the doctor in charge immediately.

In the case of subjects with adverse reactions, the safety of the subjects shall be confirmed by continuing monitoring for adverse reactions by phone call from the investigator or by visiting the subject's outpatient clinic until the symptoms are treated, and the duration shall be recorded in the case record.

12. Other matters necessary to safely and scientifically conduct clinical trials

1. Change of clinical trial protocol The purpose of the study, study design, patient population, number of subjects, and changes to the study protocol, including changes to the study procedure, and the benefits of the study, or changes to the clinical trial protocol that may affect the safety of the patient, are not official. The plan needs to be changed. These changes must be approved by the IRB prior to implementation.
2. Storage of data The head of the testing institution shall appoint a person in charge of storage for five years from the date of completion of the clinical trial, unless the retention period is specifically determined by other laws and regulations among records and data handed over from the review committee and the research manager. In addition, measures should be taken to prevent these data from being damaged or lost early due to accidents, etc.
3. Researcher's Duties

   1. Clinical trial records and supporting documents Researchers must preserve all clinical trial related documents, including all communication related to the study, patient records, consent, records of use and administration of all clinical trial drugs, and copies of case records, and ensure that these documents are not damaged or lost early due to accidents, etc. . However, after the completion of the result report (if the fact-finding investigation by the head of the Korea Food and Drug Administration is necessary, the investigation is completed), these documents must be handed over to the person in charge of storage of a separately determined testing institution.
   2. Modification of clinical trial protocol The investigator cannot modify this clinical trial protocol during the trial without the consent of the other party. If participants wish to approve a change in the clinical trial protocol, the IRB will approve the change protocol.
   3. Disclosure of data Individual patient medical information obtained as a result of this study is considered confidential, and disclosure to third parties is prohibited except as specified below. However, medical information may be provided to the patient's individual physician or other appropriate health care provider responsible for the patient's well-being. Data generated as a result of this study will be disclosed to the Institutional Review Board or regulatory authority for due diligence upon request

ELIGIBILITY:
Inclusion Criteria:

1. trainees in general surgery
2. No experience of laparoscopic cholecystectomy
3. Less than 5 experiences of laparoscopic surgery
4. Uncomplicated symptomatic gallstone disease

Exclusion Criteria:

1. Experience with laparoscopic cholecystectomy.
2. More than 5 experiences of laparoscopic surgery

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-02 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
the trainee's learning achievement | 60 days
  The Global Operative Assessment of Laparoscopic Skills, GOALS

SECONDARY OUTCOMES:
the satisfaction with the video editing method as an educational method | Participants will be followed for training period, an expected average of 60 days
  * Evaluating the anatomical structure during surgery and how difficult the surgical procedure was: a score of 10 ② Confidence in overall operation progress: evaluated on a scale of 10 ③ Value of surgical observation and video editing on the progress of the surgery: evaluated as a score of 10
postoperative complication | patients will be followed for duration of hospital stay, an expected average of 2 days
  postoperative complication : bile leakage, atelectasis, pneumonia, wound
hospital stay | patients will be followed for duration of hospital stay, an expected average of 2 days
  hospital stay(days) : The duration between the operation day and the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sung eun Park, MD, Study Director — The Catholic University of Korea
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: No